CLINICAL TRIAL: NCT04890821
Title: Early Feasibility Study (EFS) of the Cardiac Implants Percutaneous Ring Annuloplasty System for the Treatment of Functional Tricuspid Regurgitation
Brief Title: Early Feasibility Study of the Cardiac Implants Percutaneous Ring Annuloplasty System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiac Implants LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLP-100
Record Dates: First submitted 2021-05-07; First posted 2021-05-18 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Tricuspid Regurgitation Functional
Keywords: Tricuspid Valve; Annular Dilatation; Annuloplasty; Tricuspid Valve Repair

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- CI Percutaneous Ring Annuloplasty System (Experimental): Patients treated with the CI Percutaneous Ring Annuloplasty System
  Interventions: Device: CI Percutaneous Ring Annuloplasty System

INTERVENTIONS:
Device: CI Percutaneous Ring Annuloplasty System — Percutaneous transcatheter implant and adjustment of the CI ring annuloplasty system.

SUMMARY:
An early feasibility study to evaluate the safety and performance of 1) the transcatheter delivery and implantation of the Cardiac Implants (CI) annuloplasty ring and 2) the adjustment of the ring approximately 90 days following implantation in patients suffering from ≥ moderate functional tricuspid regurgitation (FTR).

DETAILED DESCRIPTION:
An early feasibility, multi-center, prospective, single-arm, non-randomized study to assess the safety and performance of the CI Percutaneous Ring Annuloplasty System in patients suffering from ≥ moderate functional tricuspid regurgitation (FTR). Additional outcomes include short and long-term changes in echocardiographic, functional, and quality of life parameters post-adjustment.

The CI Ring Annuloplasty System is a percutaneous transcatheter repair device delivered by right heart catheterization through the right internal jugular vein. The System is designed to perform annuloplasty using a Ring Delivery System (RDS) to place a complete, flexible ring over the tricuspid annulus on the atrial side of the valve. Fluoroscopy and transesophageal echocardiography are used to guide and monitor the ring placement procedure.

After implantation, the ring becomes embedded within the fibrous tissue of the tricuspid annulus. Approximately 3 months following implantation, the ring is manually adjusted under echocardiographic and fluoroscopic imaging using an Adjustment Tool (AT) until desired reduction of the tricuspid annulus dimension is achieved. Following adjustment, the AT releases a fastener, securing the ring once optimal annular reduction is achieved.

ELIGIBILITY:
Inclusion Criteria:

1. Moderate to severe functional tricuspid regurgitation (TR) defined by ASE guidelines and the European Association of Echocardiography guidelines.
2. Tricuspid valve annular diameter ≥ 40mm or > 21 mm/m2 as measured by baseline TTE in a 4-chamber view within 90 days prior to index implant procedure.
3. Age ≥ 18 years old at the time of enrollment.
4. New York Heart Associate Classification ≥ II.
5. Symptoms of right heart failure despite optimized medical therapy.
6. Multidisciplinary heart team (minimum of four physicians, including imaging, Structural Heart Disease Interventionalist, Heart Failure Cardiologist, and Cardiac Surgeon) agree that percutaneous tricuspid annuloplasty is a reasonable treatment.
7. Left Ventricular Ejection Fraction (LVEF) ≥ 30% within 90 days prior to index implant procedure
8. The subject has suitable anatomy for investigational device implantation as per imaging requirements.
9. The subject has read and signed the informed consent prior to study related procedures.
10. The subject is willing and able to comply with all required follow-up evaluations and assessments.

Exclusion Criteria:

1. Acute decompensated heart failure requiring hospital admission with 4 weeks of enrollment.
2. Severe RV dysfunction as assessed by echocardiography.
3. Primary (organic) tricuspid pathology (e.g. rheumatic, congenital, infective, etc.).
4. Currently participating in another investigational drug or device study.
5. Systolic pulmonary arterial pressure (sPAP) > 70 mmHg as measured by Transthoracic Echocardiography (TTE).
6. Subject requiring another cardiac procedure in the framework of the index procedure; subject requiring a percutaneous procedure within 30 days before or after the procedure or a cardiac surgical procedure within 3 months before or after the procedure.
7. Tricuspid valve stenosis.
8. Aortic, mitral and/or pulmonic valve stenosis and/or regurgitation more than moderate.
9. Intra-cardiac thrombus, mass or vegetation requiring active treatment.
10. Prior tricuspid repair or tricuspid replacement.
11. Known allergy to contrast media, stainless steel or nitinol that cannot be adequately pre-medicated.
12. History of cardiac transplantation.
13. Contraindication to Transthoracic/Transesophageal Echocardiography (TTE/TEE).
14. Endocarditis or severe infection within 12 months of scheduled implant procedure.
15. Myocardial Infarction (MI), percutaneous coronary intervention (PCI), or known unstable angina within the 60 days prior to the index procedure.
16. Cerebro-Vascular Accident within the previous 3 months.
17. Hemodynamic instability or on IV inotropes.
18. Contraindication to anticoagulant therapy and dual antiplatelet therapy.
19. Documented history of bleeding diathesis, hypercoagulable or active peptic ulcer or gastrointestinal bleeding within 3 months of scheduled implant procedure.
20. Severe renal impairment or on dialysis.
21. Any condition that, in the opinion of the investigator, may render the subject unable to complete the study (e.g. life expectancy < 1 year), or lead to difficulties for subject compliance with study requirements.
22. Acute anemia.
23. Chronic Oral Steroid Use ≥ 6 months.
24. Pregnant or lactating female of childbearing potential with a positive pregnancy test 24 hours before any study-related radiation exposure.
25. Pulmonary embolism within the last 6 months.
26. Tricuspid Valve Tethering distance > 10 mm.
27. Presence of transvalvular pacemaker or defibrillator leads which are determined as immobile or interfering with the procedure, as evaluated by echocardiography.
28. Inadequate TEE acoustic window for appropriate visualization of the tricuspid valve that is required for guiding the index implant procedure.
29. Contra-indicated for blood transfusion or refuses transfusion.
30. Patient undergoing emergency treatment.
31. Patient without appropriate jugular access.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Freedom from device or procedure-related mortality | 30 days post-adjustment
  Freedom from mortality determined to be primarily caused by the device or procedure in the primary endpoint cohort. Events adjudicated by a Clinical Events Committee (CEC).

SECONDARY OUTCOMES:
Safety: Incidence of device or procedure-related major adverse events (MAE) | 30, 60, and 90 days post-implant; 30 days, 3 months, 6 months, 12 months, and 2-5 years (annually) post-adjustment
  The incidence of MAEs determined to be primarily caused by the device or procedure. Events adjudicated by CEC.
Technical: Proportion of successful access, delivery, and retrieval device delivery system | 30 days post-implant and 30 days post-adjustment
  The proportion of successful access, delivery, and retrieval of the device delivery system.
Technical: Proportion of successful deployment and positioning of the ring implant. | 30 days post-implant and 30 days post-adjustment
  The proportion of successful deployment and correct/stable positioning of the ring implant.
Technical: Freedom from emergency surgery or reintervention | 30 days post-implant and 30 days post-adjustment
  The proportion of subjects free from emergency surgery or reintervention casually related to the device or access procedure.
Technical: Rate of Successful Implants | 30 days post-implant
  The proportion of subjects with successful ring implants.
Technical: Proportion of Successful Procedures | 30 days post-implant and 30 days post-adjustment
  Proportion of successful procedures, as defined in Mitral Valve Academic Research Consortium (MVARC)
Technical: Number of device stakes embedded in tissue | 30 days post-implant, 30 days post-adjustment, and 1 year post-adjustment
  Proportion of device stakes embedded in tissue vs. stakes remain embedded at follow-up, per subject, as assessed through multi-modality imaging (i.e. fluoroscopy, cine, TEE, and Cardiac CT) and evaluated by an independent Core Lab(s).
Mechanistic: Changes in TR Severity | 30 and 90 days post-implant; and 30, 90, 180, and 1-2 years (annually) post-adjustment
  The changes in TR severity, characterized per the American Society of Echocardiography (ASE) guidelines, as compared to baseline, to be evaluated by independent Core Lab.
Mechanistic: Echocardiographic changes: Changes Tricuspid Valve (TV) Annular Diameter | 30 days, 90 days, 180 days, 1 year, and 2 years post-adjustment
  Changes in TV annular diameter as compared to baseline, determined via echocardiography.
Mechanistic: Echocardiographic changes: Changes in TV Area | 30 days, 90 days, 180 days, 1 year, and 2 years post-adjustment
  Changes in TV area as compared to baseline, determined via echocardiography.
Mechanistic: Echocardiographic changes: Changes in Vena Contracta (VC) dimensions | 30 days, 90 days, 180 days, 1 year, and 2 years post-adjustment
  Changes in VC dimensions as compared to baseline, determined via echocardiography.
Mechanistic: Echocardiographic changes: Changes in Proximal isovelocity surface area (PISA) effective regurgitant orifice area (EROA) | 30 days, 90 days, 180 days, 1 year, and 2 years post-adjustment
  Changes in PISA EROA as compared to baseline, determined via echocardiography.
Mechanistic: Echocardiographic changes: Changes in Quantitive EROA | 30 days, 90 days, 180 days, 1 year, and 2 years post-adjustment
  Changes in quantitative EROA as compared to baseline, determined via echocardiography.
Mechanistic: Echocardiographic changes: Changes in TV Regurgitant Volume | 30 days, 90 days, 180 days, 1 year, and 2 years post-adjustment
  Changes in TV regurgitant volume as compared to baseline, determined via echocardiography.
Mechanistic: Echocardiographic changes: Changes in Right Atrium (RA) Dimensions | 30 days, 90 days, 180 days, 1 year, and 2 years post-adjustment
  Changes in RA dimensions as compared to baseline, determined via echocardiography.
Mechanistic: Echocardiographic changes: Changes in Right Ventricle (RV) Dimensions | 30 days, 90 days, 180 days, 1 year, and 2 years post-adjustment
  Changes in RV dimensions (cm) as compared to baseline, determined via echocardiography.
Mechanistic: Echocardiographic changes: Changes in Inferior Vena Cava (IVC) Dimensions | 30 days, 90 days, 180 days, 1 year, and 2 years post-adjustment
  Changes in IVC dimensions as compared to baseline, determined via echocardiography.
Mechanistic: Echocardiographic changes: Changes in Tricuspid Annular Plane Systolic Excursion (TAPSE) | 30 days, 90 days, 180 days, 1 year, and 2 years post-adjustment
  Changes in TAPSE as compared to baseline, determined via echocardiography.
Mechanistic: Echocardiographic changes: Changes in Left Atrium (LA) Dimensions | 30 days, 90 days, 180 days, 1 year, and 2 years post-adjustment
  Changes in LA dimensions as compared to baseline, determined via echocardiography.
Mechanistic: Echocardiographic changes: Changes in Left Ventricle (LV) Dimensions | 30 days, 90 days, 180 days, 1 year, and 2 years post-adjustment
  Changes in LV dimensions as compared to baseline, determined via echocardiography.
Functional: Changes in NYHA Classification | 1 year post-adjustment
  Changes in New York Heart Association (NYHA) classification as compared to baseline.
Functional: Changes in Distance Walked for Exercise Tolerance | 1 year post-adjustment
  Changes in distance walked, assessed by 6 Minute Walk Test
Functional: Changes in Quality of Life Scores and Sub-Domains | 1 year post-adjustment
  Changes in quality of life overall score and sub-domains in comparison to baseline values as evaluated by the Kansas City Cardiomyopathy Questionnaire (KCCQ)

OTHER OUTCOMES:
Freedom from Heart Failure Events | 30 days, 90 days, 180 days, and 1-5 years (annually) post-adjustment
  Freedom from heart failure events post-adjustment defined as a heart failure hospitalization, stratified by cardiac related vs. non-cardiac events compared to baseline.
Changes in Heart Failure Biomarkers | 180 days, 1 year, and 2 years post-adjustment
  Changes in N-terminal (NT)-pro hormone BNP (NT-proBNP) levels as compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Nodar Kipshidze, MPH, Study Director — Cardiac Implants LLC
Locations (2):
- United States (2):
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Weill Cornell Medicine-New York Presbyterian Hospital, New York, New York

IPD SHARING:
Plan to Share IPD: No